CLINICAL TRIAL: NCT04480385
Title: Study of the Technological and Operational Feasibility of a Remote Automated Monitoring System for the Post-operative Care of Surgical Patients
Brief Title: REmote Data Acquisition After SURgery
Acronym: REDASUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Rhythm Diagnostic Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-009
Record Dates: First submitted 2020-07-08; First posted 2020-07-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Visceral and Digestive Surgery
Keywords: Vital signs; Connected device; real-time monitoring; post-surgery monitoring; cardio-respiratory monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Automated Monitoring System (Experimental): MultiSense® strip will be attached on patient's thorax. The monitoring will last 7 days through post-operative monitoring room (continuous comparison with reference monitor), general ward (comparison with spot-check monitoring) and patient's home
  Interventions: Other: Remote Automated Monitoring System

INTERVENTIONS:
Other: Remote Automated Monitoring System — The patient will be monitored with conventional monitoring devices as well as the MultiSense patch

SUMMARY:
In this clinical study, the investigators will compare vital parameters measurements obtained using continuous data from reference monitors and continuous wireless MultiSense® monitoring patch in 60 patients immediately after in-ward surgery and over 7 days.

DETAILED DESCRIPTION:
The MultiSense® strip is a unique, band aid-sized, clinical signal quality, connected strip for real-time monitoring of cardio-respiratory parameters. The MultiSense® strip measures in real-time, remotely and continuously 11 clinical key-indicators by being attached to the patient thorax: Electrocardiogram (ECG) trace, heart rate, oxygen saturation, respiratory rate and relative respiration depth, pulse transit time, plethysmographic trace, perfusion index, skin temperature, physical activity and body position. Designed to be worn continuously for at least seven days, the patient can keep the patch during his sleep or in the shower.

The aim of this study is to determine the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of accuracy, connectivity, generation of artefactual data and stability of data transmission. The study population includes 60 patients undergoing visceral or digestive surgery. Once in the post-operative monitoring room, the MultiSense® strip will be attached on patient's thorax. The monitoring will last 7 days through post-operative monitoring room (continuous comparison with reference monitor), general ward (comparison with spot-check monitoring) and patient's home.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old
* Patient programmed for an elective in-ward surgery
* Patient located in Strasbourg area
* Patient with Wi-Fi and/or Cellular connectivity at home
* Patient able to receive and understand information related to the study and give written informed consent.
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient with a skin disease that would not allow the use of an adhesive
* Patient with an implantable device such as a pacemaker
* Pregnant or lactating patient
* Patient in exclusion period (determined by a previous or a current study)
* Patient under guardianship or trusteeship
* Patient under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of accuracy. | from patch placement to hospital discharge, assessed up to 1 week
  Accuracy is defined as an average measurement variation less than 3.5 percent or 5 percent of the mean value, depending on the variable with respect to the reference standard.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of connectivity. | from patch placement to hospital discharge, assessed up to 1 week
  Connectivity is defined as a time-wise ratio of missing versus total signal less than 20 percent.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of generation of artefactual data. | from patch placement to hospital discharge, assessed up to 1 week
  The generation of artefact data is defined as a percentage of outlier data less than 10 percent.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of stability of data transmission. | from patch placement to hospital discharge, assessed up to 1 week
  Data transmission stability is defined as a data transmission rate equal to or greater than 80 percent.

SECONDARY OUTCOMES:
Usability of a data acquisition patch by health care providers (HCPs) in different hospital settings assessed via questionnaires. | At hospital discharge, up to 7 days after the patch placement
  Descriptive determination of user-friendliness, comprehensibility and ease of placement, connection and removal of the data acquisition patch by healthcare providers.
User experience of surgical patients with the continuous use of a data acquisition patch during remote postoperative monitoring assessed via patient's final questionnaires. | From patch placement to its removal (7 days)
  Descriptive determination of user experience and practicalities associated with wearing the data acquisition patch (e.g. portability, duration of skin adhesion, anticipated detachment, interference with activities and stigma perception).
Assess patients' tolerability to prolonged use of an adhesive patch during remote postoperative monitoring. | From patch placement to its removal (7 days)
  Number of unexpected local and distant events attributable to the use of the adhesive data acquisition patch.

CONTACTS AND LOCATIONS:
Overall Officials: Michel VIX, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No